CLINICAL TRIAL: NCT04024852
Title: Air Pollution, Physical Activity and Cardiovascular Function of Patients With Implanted Cardioverter Defibrillators: A Randomized Controlled Trial of Indoor Versus Outdoor Activity
Brief Title: Air Pollution, Physical Activity and Cardiovascular Function of Patients With Implanted Cardioverter Defibrillators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Canada (Other Government)
Collaborators: University of Toronto (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ling Liu, Head, Air Health Effects Research Section, Health Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPAHH
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Blood Pressure
Keywords: Implanted cardioverter defibrillator; physical activity; air pollution
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants with implanted cardioverter defibrillator (ICD) were randomly divided into the control and intervention group. Both groups did daily 30-minute walked outdoors for maximum 70 days, and their data on blood pressure, pulse rate and blood oxygen saturation pre- and post-exercise were collected. Hourly ambient concentrations of PM2.5, O3, NO2, sulphur dioxide (SO2) and carbon monoxide (CO) were collected, and AQHI calculated. On days forecast with AQHI ≥5, the intervention group was advised to exercise indoors. Mixed-effects models were applied to analyze the associations between air pollution and cardiovascular measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group did daily mild exercise (walking) outdoors for 30 minutes, for maximum 70 days.
- Intervention group (Other): When Air Quality Health Index is below level 5, the intervention group did daily mild exercise (walking) outdoors for 30 minutes. When Air Quality Health Index is equal to or above level 5, the group is advised to do mild exercise indoors for 30 minutes. Total study period lasted for maximum 70 days.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — When Air Quality Health Index is below level 5, the intervention group did daily mild exercise (walking) outdoors for 30 minutes. When Air Quality Health Index is equal to or above level 5, the group is advised to do mild exercise indoors for 30 minutes.
  Arms: Intervention group

SUMMARY:
This study investigated whether patients with an implanted cardioverter defibrillator (ICD) who followed advice to exercise indoors on high air pollution days had reduced adverse impacts on cardiovascular measures compared with those who exercised outdoors on those days. Participants were randomly divided into the control and intervention groups. Both groups walked for 30 minutes outdoors every day for maximum 70 days, and their blood pressure, pulse rate and blood oxygen saturation pre- and post-exercise were measured. Hourly ambient concentrations of air pollutants were collected. On days forecast with Air Quality Health Index was equal to or higher than 5, the intervention group was advised to exercise indoors.

DETAILED DESCRIPTION:
Background: The Air Quality Health Index (AQHI) is a risk communication tool intended to provide information to the public on current and forecast air quality conditions. It was developed by the Canadian government to help the public make decisions to limit short-term exposure to air pollution and adjust their activity when air pollution levels are high, particularly for people who are sensitive to air pollution. Little research has been done to characterize the benefits of following AQHI advice. The AQHI is based on a weighted sum of concentrations of nitrogen dioxide (NO2), ozone (O3), and particulate matter of median aerodynamic diameter ≤ 2.5 µm (PM2.5) to provide information to the public on current and forecasted air quality conditions.

Objective: This study investigated whether patients with an implanted cardioverter defibrillator (ICD) who followed advice to exercise indoors on high AQHI days had reduced adverse impacts on cardiovascular measures compared with those who exercised outdoors on those days.

Methods: Participants with ICD were randomly divided into the control and intervention group. Both groups did daily 30-minute walked outdoors for maximum 70 days, and their data on blood pressure, pulse rate and blood oxygen saturation pre- and post-exercise were collected. Hourly ambient concentrations of PM2.5, O3, NO2, sulphur dioxide (SO2) and carbon monoxide (CO) were collected, and AQHI calculated. On days forecast with AQHI ≥5, the intervention group was advised to exercise indoors. Mixed-effects models were applied to analyze the associations between air pollution and cardiovascular measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with structural heart disease with an implanted cardioverter difribrillator (ICD) in situ
* 18 years of age and older
* living and working in Toronto (Canada) and surrounding area
* The participants are healthy enough for mild outdoor activity (a 30-minute walk).

Exclusion Criteria:

* Decompensated heart failure (CHF) patients defined as a hospital admission for CHF or intravenous ionotropic administration within the preceding 6 months
* patients on class 1 and 11 antiarrhythmics and congenital heart disease patients
* patients who have experienced frequent or recent shocks (within the last 3 months of the experiment)
* patients who have underlying conditions that would interfere with mild daily exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
blood pressure | before and after 30-minute exercise
  Systolic and diastolic blood pressure is measured in the dominant arm with the subject seated, using an automated sphygmomanometer (BIOS Medical, Newmarket, Ontario, Canada), taking the average of the three readings one minute apart
pulse rate | before and after 30-minute exercise
  Pulse rate is measured using the pulse oximeter.
blood oxygen saturation | before and after 30-minute exercise
  Oxygen saturation is measured using a pulse oximeter with a finger sensor (Choice MMed, Beijing Choice Electronic, China). The oximeter is run continuously for 3 minutes to obtain each measurement and the average oxygen saturation during this period is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, MD, PHD, Principal Investigator — Health Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu L, Urch B, Nanthakumar K, Chen L, Smith-Doiron M, Brook JR, Speck M, Silverman F, Stieb DM. Air Pollution, Physical Activity, and Cardiovascular Function of Patients With Implanted Cardioverter Defibrillators: A Randomized Controlled Trial of Indoor Versus Outdoor Activity. J Occup Environ Med. 2020 Apr;62(4):263-271. doi: 10.1097/JOM.0000000000001795. PMID 31880734